CLINICAL TRIAL: NCT04000334
Title: Early Transcranial Doppler Goal Directed Therapy After Cardiac Arrest: a Pilot Study
Acronym: GOODYEAR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the difficulty of recruiting patients and the fact that, despite the team's best efforts, the inclusion period initially planned had largely passed, it did not appear ethical to continue the study.
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHM-2019/S3/04
Record Dates: First submitted 2019-06-22; First posted 2019-06-27 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Arrest; Cerebral Lesion; Ischemic Encephalopathy; Ischemic Reperfusion Injury
Keywords: cardiac arrest; cerebral blood flow; cerebral autoregulation; transcranial doppler
MeSH Terms: conditions — Heart Arrest; Brain Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cerebral hypoperfusion (group A) (Experimental): Cerebral hypoperfusion will be defined by an abnormal TCD at inclusion (t0) when two of the three measured values are abnormal using the following thresholds: Vm < 30 cm/s, Vd < 20 cm/s, PI > 1.4.
  Interventions: Other: MAP increased to optimize cerebral blood flow
- Normal cerebral perfusion (group B) (Active Comparator): Normal cerebral perfusion will be defined by a normal TCD at inclusion (t0) when two of the three measured values are normal using the following thresholds: Vm > 30 cm/s, Vd > 20 cm/s, PI < 1.4.
  Interventions: Other: MAP between 65 and 85 mmHg

INTERVENTIONS:
Other: MAP increased to optimize cerebral blood flow — MAP will be increased to 90-100 mmHg with norepinephrine. If TCD is still abnormal with a MAP of 90-100 mmHg, MAP will be increased to 100-110 mmHg. At each step, all CBF determinants will be recorded as well as cardiac output and Veinous jugular oxygen saturation (SvjO2). When TCD is normalized with no complications, MAP will be maintained at 90-100 or 100-110 mmHg during 24 hours.
  Arms: Cerebral hypoperfusion (group A)
Other: MAP between 65 and 85 mmHg — MAP will be maintained between 65-85 mmHg, using a norepinephrine infusion as needed.
  Arms: Normal cerebral perfusion (group B)

SUMMARY:
Hypoxic-ischaemic brain injury (HIBI) is the main cause of death in patients who are comatose after resuscitation from cardiac arrest. Current guidelines recommend to target a mean arterial pressure (MAP) above 65 mmHg to achieve an adequate organ perfusion. Moreover, after cardiac arrest, cerebral autoregulation is dysregulated and cerebral blood flow (CBF) depends on the MAP. A higher blood pressure target could improve cerebral perfusion and HIBI. Transcranial Doppler (TCD) is a non-invasive method to study CBF and its variations induced by MAP.

The aim of this study is to test the feasibility of an early-goal directed hemodynamic management with TCD during the first 12 hours after return of spontaneous circulation (ROSC).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in the Intensive Care Unit (ICU) under mechanical ventilation with a Glasgow Coma Scale ≤ 8/15 after in- or out-of-hospital cardiac arrest
* Mean arterial pressure between 65 and 85 mmHg with or without vasopressor support

Exclusion Criteria:

* Age < 18 years old
* No flow (time between cardiac arrest and the beginning of cardiac massage) > 15 minutes or unknown
* Low flow ((time between cardiac arrest and ROSC: return of spontaneous circulation)> 60 minutes
* Time between ROSC and inclusion > 12 hours
* Transcranial doppler unavailable
* Cardiac arrythmia
* Patient under extracorporeal life support before inclusion or at risk of being referred for assistance due to cardiogenic shock with high dose of vasopressors before inclusion (MAP < 65 mmHg with norepinephrine or epinephrine > 1 µg/kg/min or dobutamine > 10 µg/kg/min)
* Severe cardiac dysfunction defined by left ventricular ejection fraction < 20% or aortic Velocity Time Integral (VTI: measured with trans-thoracic echocardiography) < 14 cm with dobutamine > 10µg/kg/min
* Patient under Extracorporeal Membrane Oxygenation (ECMO) for Acute Respiratory Distress Syndrome (ARDS) before inclusion
* Cardiac arrest secondary to brain injury such as stroke, subarachnoid hemorrhage or traumatic brain injury
* Hemorrhagic shock
* Any acute pathology that requires strict blood pressure control (aortic dissection, stroke, cardiogenic pulmonary edema with high blood pressure)
* Decision of withdrawing or withholding life sustaining treatment before inclusion or considered during the first 12 hours of ICU management
* Patient with a modified Rankin scale (MRS) 4 or 5 prior to resuscitation
* Pregnancy or lactation
* Patients already enrolled in another clinical study on cardiac arrest
* Patients with judicial protection
* No social security coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2023-07-08 (Actual); Study Completion 2023-07-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in whom the transcranial doppler goal directed therapy will result in a modification of MAP targets | In the first hour after inclusion
  Proportion of patients in whom transcranial doppler goal directed therapy will result in a modification of MAP targets.

SECONDARY OUTCOMES:
Cerebral blood flow modifications induced by increasing MAP | At the 6th, 12th, 24th, 48th and 72nd hour after inclusion
  Transcranial doppler data modifications induced by increasing MAP to 90-100 mmHg and 100-110 mmHg.
Cerebral oxygenation modifications induced by increasing MAP | At the 6th, 12th, 24th, 48th and 72nd hour after inclusion
  Bulb jugular venous oxygen saturation modifications induced by increasing MAP at 90-100 mmHg and 100-110 mmHg.
Undesirable events induced by increasing MAP | At te 24th hour after inclusion
  Number of cardiovascular events defined by new onset of severe cardiac arrythmias, acute coronary syndromes, cardiogenic pulmonary edema, cardiogenic shock or cardiac arrest
Undesirable events induced by increasing MAP | At the 72nd hour after inclusion
  Number of neurologic events defined by intracranial hematoma or brain death
Plasmatic concentrations of Neuron Specific Enolase | At the 72nd hour after inclusion
  Neuron Specific Enolase (NSE) plasmatic concentrations at H+72h after cardiac arrest
28 day survival | 28 days after inclusion
  Proportion of patients alive 28 days after inclusion
90 days survival | 90 days after inclusion
  Proportion of patients alive 90 days after inclusion
Measure of the degree of disability in the activities of daily living of the included patients | 90 days after inclusion
  Modified Rankin scale (MRS) 90 days after inclusion. The scale runs from 0-6, running from perfect health without symptoms to death.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Chudeau, MD, Principal Investigator — Centre Hospitalier Le Mans, Intensive Care Unit
Locations (1):
- Centre Hospitalier Le Mans, Le Mans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meunier J, Engrand N, Saulnier P, Deye N, Landais M, Cariou A, Guitton C, Chudeau N. Transcranial Doppler goal-directed therapy after cardiac arrest (GOODYEAR): a feasibility study. Resusc Plus. 2025 Jun 14;25:101001. doi: 10.1016/j.resplu.2025.101001. eCollection 2025 Sep. PMID 40677967